CLINICAL TRIAL: NCT06543862
Title: Autonomous Artificial Intelligence Versus AI Assisted Human Optical Diagnosis of Colorectal Polyps
Brief Title: Autonomous Artificial Intelligence Versus AI Assisted Human Optical Diagnosis
Acronym: CADx-Prosp
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Daniel Von Renteln, Principal Investigator, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-12306
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Colonic Polyp; Artificial Intelligence
Keywords: optical diagnosis, artificial intelligence
MeSH Terms: conditions — Colonic Polyps | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): The endoscopist will make an optical diagnosis (OD) prediction for all small polyps (up to 10 mm) in white light (WL). Then, the endoscopist will make another OD prediction using image enhanced endoscopy (IEE) modes. After that, CADx will be activated in the IEE mode and a CADx prediction will be documented. Finally, after seeing the CADx prediction, the endoscopist will make a final prediction, which can agree or disagree with the autonomous CADx one. Polyps will be resected and sent to a pathology lab, where a pathologic diagnosis (blinded to the endoscopist's predictions) will be rendered.
  Interventions: Other: CADx (AI) system

INTERVENTIONS:
Other: CADx (AI) system — The CADx system will be used to predict the histopathology of the polyp detected.

SUMMARY:
Computer-aided image-enhanced endoscopy can predict the nature of colorectal polyps with over 90% accuracy. This technology uses artificial intelligence (AI) to analyze video recordings of polyps, learning to make diagnoses in real-time. This means that doctors can get immediate predictions about small polyps during the procedure, reducing the need for separate pathology exams and saving costs, ultimately improving patient care.

Human and AI interactions are complex and a framework to reap synergistic effects CADx systems when used by humans to harness optimal performance needs to be established. AI solutions in medicine are usually developed to be used as assistive devices, however, then they rely on humans to correct AI errors. Optical polyp diagnosis is a complex task. Non experts usually achieve diagnostic accuracy in 70-80%. CADx systems have a similar diagnostic accuracy when used autonomously. Clinical evaluation of CADx systems showed that CADx assisted OD performs equally to the operator performance when using non CADx assisted OD. To harness a benefit of clinical CADx implementation we would have to find a way that synergies between human and CADx come into play to eliminate cases in which CADx assisted and/ or human OD results in low diagnostic accuracy and also addresses the problem of serrated polyp recognition.

DETAILED DESCRIPTION:
Our study hypothesis is that for CADx implementation, instead of using the high/low confidence framework, identifying cases with suboptimal diagnostic accuracy could be facilitated through identifying cases in which CADx and endoscopist disagreed in their diagnosis. Eliminating such cases might separate out cases with low accuracy when using CADx assisted OD. Since endoscopists have a high sensitivity but low specificity for serrated polyp OD, this framework will also allow us to implement a strategy to adequately manage serrated polyps found in the cohort.

ELIGIBILITY:
Inclusion Criteria:

* Indication for full colonoscopy.

Exclusion Criteria:

* Known inflammatory bowel disease
* Active colitis
* coagulopathy
* familial polyposis syndrome
* poor general health, defined as an American Society of Anesthesiologists class >3
* emergency colonoscopy

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of optical diagnosis, for polyps 1-5mm, compared with an agreed upon CADx-assisted diagnosis | up to 100 weeks
  Accuracy of optical diagnosis, for polyps 1-5mm, compared with an agreed upon CADx-assisted diagnosis , when histopathology results are used as the reference

SECONDARY OUTCOMES:
Accuracy of optical diagnosis, for polyps 1-10mm, compared with an agreed upon CADx-assisted diagnosis | up to 100 weeks
  Accuracy of optical diagnosis, for polyps 1-10mm, compared with an agreed upon CADx-assisted diagnosis, when histopathology results are used as the reference
Test characteristics, including recall, specificity, positive and negative predictive values (PPV/NPV), and particularly the NPV of rectosigmoid neoplastic polyps. | up to 100 weeks
  A ≥90% NPV will be used as a quality benchmark for a strategy to not resect such diminutive polyps.
Agreement of surveillance interval recommendations of AI-A and AI-H compared with the pathology-based recommendations | up to 100 weeks
  For surveillance interval assignment, the pathology results of concomitant polyps >5 mm (including multiple concomitant polyps of all sizes and histology) will be considered when calculating the surveillance interval recommendation. Surveillance recommendations will be based on the 2020 United States Multi Society Task Force Guidelines as is current standard of practice at our center.
Proportion of patients for whom an immediate surveillance recommendation can be directly provided for each approach, and how often histopathology-based polyp examination would have been avoided. | up to 100 weeks
  The potential cost-effectiveness of OD (either approaches) will be evaluated using the measured described above.
Variability of OD (AI-A and AI-H) across participating endoscopists. | up to 100 weeks
  Each participating endoscopist will conduct a similar number of optical diagnoses to assess endoscopist-related factors.
Cost-effectiveness of OD ((AI-A and AI-H) | up to 100 weeks
  A cost-effectiveness model will be applied to better quantify costs and understand cost impact including key cost drivers when generalized to a broader screening population.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, MD, Principal Investigator — University of Montreal Medical Center (CHUM)
Locations (1):
- Ghislaine Ahoua, Montreal, Quebec, Canada